CLINICAL TRIAL: NCT01566383
Title: Assessing Normal Multichannel Intraluminal Impedance (MII)-pH Parameters for Today's Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to meet recruitment goals
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Medical Director, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 120288
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Identify Normal MII-pH Parameters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Healthy volunteers who are matched (age, weight, gender) to the general patient population undergoing manometry and pH monitoring for GERD will undergo the same procedures to determine pH levels in people without reflux symptoms as compared to pH levels in those patients who have been diagnosed with reflux.
  Interventions: Procedure: 24-hr pH monitoring

INTERVENTIONS:
Procedure: 24-hr pH monitoring — Visit 1
  The following will be done:
  * A medical history including review of your current drugs;
  * Collection of demographic information;
  * A manometry, before the 24-hour pH testing, to find the junction between the esophagus and stomach;
  * 24-hour pH testing will be done
  Visit 2
  You will return to the clinic 24 hours after the visit 1 and the following will occur:
  * The catheter will be removed from your nose; and
  * You will return the recording device

SUMMARY:
The normal values of a Multichannel Intraluminal Impedance (MII)-pH study can vary between ages, gender, race and different values of body mass index (BMI). This fact can cause new modifications in the normal values such as making new scales for different age groups or BMI groups.

Our aim is to find the normal esophageal MII-pH parameter ranges in volunteers who never experienced reflux related symptoms and are in between the same ranges of age and BMI of our gastroesophageal reflux disease (GERD) patient population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between the ages of 33-65
* BMI range of 23.9 - 38.9
* Ability to give consent to participate in study

Exclusion Criteria:

* History of extraesophageal reflux disease symptoms such as chronic or acute cough and/or throat clearing and /or non-cardiac chest pain.
* History of gastroesophageal reflux disease (GERD) such as heartburn and/or regurgitation.
* History of proton pump inhibitor (PPI) usage ten days prior to the procedure (MII-pH) or H2RA's two days prior to MII-pH and antacids usage on the procedure day.
* History of thoracic, gastric or esophageal surgery.
* Histories of Diabetes Mellitus, neurological disorders, gastrointestinal disease, taking medication that alter the intragastric acidity or esophageal motility.
* Pregnancy or nursing mothers.
* Alcohol consumption >40g/day, smoking >10cigarettes/day.

Ages: 33 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08-27 (Actual); Study Completion 2013-08-27 (Actual)

PRIMARY OUTCOMES:
Identify normal esophageal MII-pH parameter ranges in healthy volunteers | Following 24-hr pH monitoring
  Our aim is to find the normal esophageal MII-pH parameter ranges in volunteers who never experienced reflux related symptoms and are in between the same ranges of age and BMI of our GERD patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Vaezi, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No